CLINICAL TRIAL: NCT06637332
Title: DAPTO-SNAP: Daptomycin vs. Vancomycin for the Treatment of Methicillin Resistant S. Aureus Bacteremia
Brief Title: Daptomycin vs. Vancomycin for the Treatment of Methicillin Resistant S. Aureus Bacteremia
Acronym: DAPTO-SNAP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Todd C. Lee MD MPH FIDSA (Other)
Collaborators: University of Melbourne (Other); The Peter Doherty Institute for Infection and Immunity (Other)
Responsible Party: Sponsor-Investigator, Todd C. Lee MD MPH FIDSA, Associate Professor of Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-10666; 466322 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Staphylococcus Aureus Septicemia; Staphylococcus Aureus Bacteremia; S. Aureus Bacteremia; S. Aureus Bloodstream Infection; Staphylococcus Aureus Endocarditis
Keywords: S. aureus bacteremia; Methicllin resistant; MRSA; S. aureus bloodstream infection; Daptomycin; Vancomycin
MeSH Terms: interventions — Daptomycin; Injections; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daptomycin (Experimental): Daptomycin given by injection at a dose determined by the treating clinicians but no less than 6mg/kg
  Interventions: Drug: Daptomycin for Injection
- Vancomycin (Active Comparator): Vancomycin given by injection at a dose determined by the treating clinicians to achieve a trough-based or AUC-based target
  Interventions: Drug: Vancomycin (IV)

INTERVENTIONS:
Drug: Daptomycin for Injection — Daptomycin given by injection at a dose determined by the treating team but not to be less than 6mg/kg
  Arms: Daptomycin
Drug: Vancomycin (IV) — Vancomycin by injection to be given at a dose selected by the treating team to achieve a desired trough level or AUC-based target, as determined by local standards of care
  Arms: Vancomycin

SUMMARY:
This is an open label randomized controlled trial for patients with methicillin resistant S. aureus (MRSA) bloodstream infection which will directly compare the two most commonly used therapies, vancomycin and daptomycin.

This study is an approved sub-study of The Staphylococcus aureus Network Adaptive Platform (SNAP) trial (NCT05137119)

ELIGIBILITY:
The participant must meet all inclusion and exclusion criteria for the SNAP Platform (NCT05137119) and also the following inclusion and exclusion criteria:

Inclusion Criteria:

* Methicillin-resistant S. aureus bacteremia

Exclusion Criteria:

* Severe allergy or non-severe rash to vancomycin or daptomycin
* Suspected or confirmed MRSA pneumonia
* Known vancomycin minimum inhibitory concentration (MIC) greater than or equal to 2mg/L or daptomycin MIC greater than or equal to 1mg/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Desirability of Outcome Ranking (DOOR) | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  Desirability of Outcome Ranking (DOOR) - an ordinal outcome with 5 levels defined:
  Rank 1 - Alive without complication Rank 2 - Alive with 1 complication Rank 3 - Alive with 2 complications Rank 4 - Alive with 3 complications Rank 5 - Dead
  Complications include:
  1. Clinical failure: Absence of resolution of clinical signs and symptoms of S. aureus bacteremia such that no additional antibiotic therapy is required or anticipated.
  2. Infectious Complications: Including new endocarditis; new evidence of other deep metastatic foci (e.g., osteomyelitis or deep abscess); relapse of MRSA bacteremia after a patient has sterilized their initial blood cultures; readmission for subsequent care of S. aureus bacteremia; need for unplanned source control procedures; change of therapy due to inadequate clinical response.
  3. Serious adverse drug event (Common Terminology Criteria class 4) due to study drug OR adverse drug event (classes 1-3) leading to discontinuation of the study drug

SECONDARY OUTCOMES:
Clinical failure | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  Defined as the absence of resolution of clinical signs and symptoms of S. aureus bacteremia such that no additional antibiotic therapy is required or anticipated for its treatment.
Serious Adverse Event or Adverse Event Leading to Discontinuation | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  Defined as a serious adverse drug event (Common Terminology Criteria for Adverse Events (CTCAE) class 4) presumed due to study drug OR adverse drug event (CTCAE classes 1-3) leading to discontinuation of the study drug
All cause mortality | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  Death from any cause
Infectious Complications | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  Defined as change in therapy for inadequate clinical response; new endocarditis; new evidence of other deep metastatic foci (e.g., osteomyelitis or deep abscess); relapse of MRSA bacteremia after a patient has sterilized their initial blood cultures; readmission for subsequent care of S. aureus bacteremia; need for unplanned source control procedures; change of antibiotic therapy due to inadequate clinical response.
  New implies that the complication was not suspected at enrollment and is not a function of delay to diagnostic testing.
Drug Induced Myostitis | Occurring while on therapy up to day 42 from enrollment in SNAP (NCT05137119)
  Defined as a creatinine kinase level greater than or equal to 5 times the upper limit of normal
Eosinophilic pneumonia | Occurring while on therapy up to day 42 from enrollment in SNAP (NCT05137119)
  Defined as the development of symptomatic eosinophilic pneumonia as diagnosed by the treating team in consultation with the appropriate specialists

CONTACTS AND LOCATIONS:
Overall Officials: Todd C Lee, MD MPH FIDSA, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (13):
- Australia (10):
  - Concord Repatriation and General Hospital, Concord, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Campus (Monash Medical Centre + Jesse McPherson Private Hospital), Clayton, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Canada (3):
  - Fraser Health Authority (Surrey Memorial Hospital), Surrey, British Columbia
  - Newfoundland Health Services (Health Sciences Centre and St. Clare's Mercy Hospital), St. John's, Newfoundland and Labrador
  - McGill University Health Centre (Royal Victoria Hospital and Montreal General Hospital), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing policies are dependent on the policies of the SNAP Platform (NCT05137119)

REFERENCES:
- [Background] Zhang G, Zhang N, Xu J, Yang T, Yin H, Cai Y. Efficacy and safety of vancomycin for the treatment of Staphylococcus aureus bacteraemia: a systematic review and meta-analysis. Int J Antimicrob Agents. 2023 Oct;62(4):106946. doi: 10.1016/j.ijantimicag.2023.106946. Epub 2023 Aug 4. PMID 37543121
- [Background] Fowler VG Jr, Boucher HW, Corey GR, Abrutyn E, Karchmer AW, Rupp ME, Levine DP, Chambers HF, Tally FP, Vigliani GA, Cabell CH, Link AS, DeMeyer I, Filler SG, Zervos M, Cook P, Parsonnet J, Bernstein JM, Price CS, Forrest GN, Fatkenheuer G, Gareca M, Rehm SJ, Brodt HR, Tice A, Cosgrove SE; S. aureus Endocarditis and Bacteremia Study Group. Daptomycin versus standard therapy for bacteremia and endocarditis caused by Staphylococcus aureus. N Engl J Med. 2006 Aug 17;355(7):653-65. doi: 10.1056/NEJMoa053783. PMID 16914701